CLINICAL TRIAL: NCT03436641
Title: Study of Microcirculation in Cardiogenic Shock
Brief Title: Microcirculation in Cardiogenic Shock
Acronym: MicroShock
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6951
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Cardiogenic shock is usually defined as primary cardiac dysfunction with low cardiac output leading to critical organ hypo perfusion and tissue hypoxia. Despite progress in the management of cardiogenic shock, mortality remains unacceptably high.

This significant mortality, close to 40 %, is partly due to profound alterations of microcirculatory blood flow in cardiogenic shock, leading to multi organ failure, despite restoration of macro-hemodynamic parameters such as blood pressure and cardiac output. The microcirculation is the terminal vascular network of the systemic circulation consisting of microvessels with diameters < 20 μm including arterioles, capillaries, and venules. This part of the circulation is critical as it is responsible for nutrient delivering and oxygen transfer from the erythrocytes in the capillaries to the parenchymal cells to meet their metabolic demands, but it is also the area where water, other gases, hormones and waste products are exchanged.

Hence, the evaluation of clinical signs of peripheral hypoperfusion reflecting microvascular perfusion is of interest. We aimed to study these parameters such as skin capillary refill time (CRT), mottling and central-to-toe temperature difference (ΔTc-p) in a cardiogenic shock population. Assessing the prognosis of these microcirculation parameters and their interaction with macrocirculation parameters such as arterial pressure, cardiac index, left ventricular ejection fraction is also the aim of this study. Lastly, looking at the prognostic value of these markers seems interesting.

ELIGIBILITY:
Inclusion Criteria:

* major patient (≥18 years old)
* Patient with a cardiogenic shock table defined by the association of low cardiac output even though the filling pressures are normal or high, causing hypoperfusion and organ pain
* patient affiliated to a social security scheme
* patient (or family member / trusted or close) who has agreed to participate in the study

Exclusion Criteria:

* refusal of the patient to participate in the study
* patients with dark skin preventing the evaluation of clinical markers of microcirculation.
* subject under the protection of justice
* subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Standard management of cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
incidence of microcirculatory impairment in cardiogenic shock | 28 days
  evaluate the incidence of clinical parameters of involvement of microcirculation in cardiogenic shock, and their prognosis in the outcome of these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid MERDJI, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - CHU Nancy - Hôpital Brabois, Nancy
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided